CLINICAL TRIAL: NCT05380206
Title: Functional Knee Phenotypes of Patients Operated on for Total Knee Arthroplasty. Comparison With a Reference Non Arthritic Population
Brief Title: Functional Knee Phenotypes of Patients Operated on for Total Knee Arthroplasty
Acronym: FP-Knee
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8193
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee; Osteoarthritis; Knee osteoarthritis; knee arthroplasty; Total knee arthroplasty; Navigated implantation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to analyze the coronal alignment of a large population of patients undergoing total knee arthroplasty using a modern classification of the knee phenotypes found in a population of non-osteoarthritic patients.

DETAILED DESCRIPTION:
Methods Five hundred and four navigated total knee arthroplasties will be analyzed. The following angles will be measured with a computer image free navigation system: medial femorotibial mechanical angle without stress and with maximum manual stress to reduce deformation, and medial distal femoral mechanical angle. The native medial distal femoral and medial proximal tibial angles will be calculated. The data will be analyzed as numerical and categorical data. These data will be then compared with those published in a non-arthritic population, considered as a control group.

The main criterion will be the percentage of subjects with normal overall coronal alignment, defined by the association of a normal native medial distal femoral angle and a normal native medial proximal tibial angle. The secondary criteria will be the percentages of subjects with normal medial femorotibial mechanical angle, normal native medial distal femoral angle and normal native medial proximal tibial angle. The influence of gender on primary and secondary criteria in the study group will be analyzed. The most frequent phenotypes in the study group will be identified.

ELIGIBILITY:
Inclusion criteria:

* Patient aged ≥ 18 years
* Patient operated between 01/01/2011 to 02/28/2021 by two experienced surgeons of a total knee prosthesis using a navigation system without image (OrthoPilot ®, Aesculap, Tuttlingen, FRG) allowing to measure during the intervention the anatomical parameters of the subject before implantation;
* Records including a complete intraoperative anatomical analysis;
* Subject who has not expressed his opposition, after being informed, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Impossibility of giving the subject informed information (difficulties in understanding the subject, etc.)
* Incomplete or absent anatomical analysis
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient aged ≥ 18 years operated between 01/01/2011 to 02/28/2021 by two experienced surgeons of a total knee prosthesis using a navigation system without image (OrthoPilot ®, Aesculap, Tuttlingen, FRG) allowing to measure during the intervention the anatomical parameters of the subject before implantation;
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with normal overall coronal alignment, defined by the association of a normal native medial distal femoral angle and a normal native medial proximal tibial angle | Files analysed retrospectively from January 01, 2011 to February 28, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, PhD, Principal Investigator — Service de Chirurgie Orthopédique Pédiatrique - CHU de Strasbourg - France
Locations (1):
- Service de Chirurgie Orthopédique Pédiatrique - CHU de Strasbourg - France, Strasbourg, France